CLINICAL TRIAL: NCT06634797
Title: A Phase 4, Randomized, Observer-blind, Placebo-controlled, Crossover Study to Assess Cardiac Troponin Levels After mRNA-1273.712 Vaccine in Participants 12 Through 30 Years of Age
Brief Title: A Study to Investigate Cardiac Troponin Levels After mRNA-1273.712 Vaccine in Participants 12 Through 30 Years of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: mRNA-1273-P404
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
Keywords: mRNA-1273.712; Vaccine; Cardiac Troponin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: mRNA-1273.712 then Placebo (Experimental): Participants will receive mRNA-1273.712 followed by placebo 28 days later.
  Interventions: Biological: mRNA-1273.712; Biological: Placebo
- Sequence 2: Placebo then mRNA-1273.712 (Experimental): Participants will receive placebo followed by mRNA-1273.712 28 days later.
  Interventions: Biological: mRNA-1273.712; Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1273.712 — Intramuscular (IM) injection.
Biological: Placebo — Sodium chloride for IM injection.

SUMMARY:
The primary objective of this study is to assess cardiac troponin I (cTnI) values in participants who received mRNA-1273.712 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Investigator's assessment that participant understands and is willing and physically able to comply with protocol-mandated follow-up, including all procedures.
2. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).
3. Contraceptive use by participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

1. History of anaphylaxis or severe hypersensitivity reaction requiring medical intervention after receipt of any mRNA vaccine or therapeutic or any components of an mRNA vaccine or therapeutic.
2. Has known history of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 3 months prior to enrollment.
3. Has a documented history of myocarditis or pericarditis.
4. Is acutely ill or febrile (temperature ≥38.0 degrees Celsius [°C]/100.4 degrees Fahrenheit [°F]) less than 72 hours prior to or at the Screening Visit or Day 1.
5. Has known conditions that may cause elevated cTnI.

   * Cardiac disease/conditions including rhythm disorders and congenital heart disease
   * Diabetes
   * Uncontrolled hypertension (defined as systolic blood pressure >140 millimeter of mercury (mmHg) or diastolic blood pressure >90 mmHg)
   * Alcohol or substance abuse
   * Kidney disease
   * Severe obesity, defined as body mass index (BMI) ≥40 kilograms per square meter (kg/m^2) (>20 years) or severe obesity defined as BMI for sex and age ≥120% of the 95th percentile [BMI ≥35 kg/m^2] (for 12 to 20 years)
6. Currently has symptomatic acute or unstable chronic disease requiring medical or surgical care, to include significant change in therapy or hospitalization for worsening disease, at the discretion of the Investigator.
7. Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation, or that could interfere with safety assessments or interpretation of results according to the Investigator's judgment.
8. Reported history of congenital or acquired immunodeficiency (eg, human immunodeficiency virus [HIV]), immunosuppressive condition or immune-mediated disease, asplenia, or recurrent severe infections disease.
9. History of Guillain-Barré syndrome.
10. Receipt of the following:

    * Coronavirus disease 2019 (COVID-19) vaccine within 3 months prior to the first injection or if planning to receive at any time during the study (except for study intervention).
    * Any other licensed vaccine within 28 days before the study injection or planned receipt prior to end of study (EOS).
    * Systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screening (for corticosteroids ≥10 milligrams (mg)/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
    * Systemic immunoglobulins or blood products within 3 months prior to the Screening/Baseline Visit or plans for receipt during the study.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Velocity Clinical Research, Phoenix, Phoenix, Arizona
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Velocity Clinical Research, Banning, San Bernardino, California
  - Velocity Clinical Research, Washington DC, Washington D.C., District of Columbia
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - Velocity Clinical Research, Boise, Meridian, Idaho
  - Velocity Clinical Research, Valparaiso, Valparaiso, Indiana
  - Velocity Clinical Research, Covington, Covington, Louisiana
  - Velocity Clinical Research, Lafayette, Lafayette, Louisiana
  - Velocity Clinical Research, New Orleans, New Orleans, Louisiana
  - Velocity Clinical Research, Gulfport, Gulfport, Mississippi
  - Velocity Clinical Research, Grand Island, Grand Island, Nebraska
  - Velocity Clinical Research, Lincoln, Lincoln, Nebraska
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Velocity Clinical Research, Albuquerque, Albuquerque, New Mexico
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - Velocity Clinical Research, Durham, Durham, North Carolina
  - Velocity Clinical Research, Cleveland, Beachwood, Ohio
  - Velocity Clinical Research, Cincinnati, Blue Ash, Blue Ash, Ohio
  - Velocity Clinical Research, Cincinnati, Cincinnati, Ohio
  - Velocity Clinical Research, Anderson, Anderson, South Carolina
  - Velocity Clinical Research, Abilene, Abilene, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio (500 participants in each injection sequence) to receive 2 study injections (mRNA-1273.712 and placebo) in a crossover design.
Groups:
- Sequence 1: mRNA-1273.712 Then Placebo: Participants received mRNA-1273.712 as an intramuscular (IM) injection on Day 1 of the study. Participants then received placebo matched to mRNA-1273.712 as an IM injection on Day 29 of the study.
- Sequence 2: Placebo Then mRNA-1273.712: Participants received placebo matched to mRNA-1273.712 as an IM injection on Day 1 of the study. Participants then received mRNA-1273.712 as an IM injection on Day 29 of the study.
Period: Overall Study
Arm/Group | Sequence 1: mRNA-1273.712 Then Placebo | Sequence 2: Placebo Then mRNA-1273.712
Started | 500 | 500
Received Study Vaccination | 500 | 497
Completed | 438 | 424
Not Completed | 62 | 76
Not completed — Other Than Specified | 1 | 1
Not completed — Withdrawal by Subject | 12 | 21
Not completed — Physician Decision | 3 | 3
Not completed — Lost to Follow-up | 46 | 48
Not completed — Adverse Event | 0 | 1
Not completed — Screen Failure | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomization Set: Included all participants who were randomized in the study.
Groups:
- Sequence 1: mRNA-1273.712 Then Placebo: Participants received mRNA-1273.712 as an IM injection on Day 1 of the study. Participants then received placebo matched to mRNA-1273.712 as an IM injection on Day 29 of the study.
- Total: Total of all reporting groups
Arm/Group | Sequence 1: mRNA-1273.712 Then Placebo | Sequence 2: Placebo Then mRNA-1273.712 | Total
Number analyzed (Participants) | 500 | 500 | 1000
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.7 (5.73) | 20.0 (5.71) | 19.8 (5.72)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 235 | 215 | 450
  Adults (18-64 years) | 265 | 285 | 550
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 266 | 272 | 538
  Male | 234 | 228 | 462
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 68 | 79 | 147
  Not Hispanic or Latino | 423 | 417 | 840
  Unknown or Not Reported | 9 | 4 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 320 | 334 | 654
  Black or African American | 132 | 108 | 240
  Asian | 19 | 14 | 33
  American Indian or Alaska Native | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Multiple | 21 | 30 | 51
  Other | 3 | 7 | 10
  Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Elevated Cardiac Troponin I (cTnI) at Day 4 or Day 32 (3 Days After Injection 1 or Injection 2)
Description: Elevated cTnI was defined as >53.53 picograms per milliliter (pg/mL) in males and >38.64 pg/mL in females.
  One participant who was included in the analysis, had an elevation of cTnI pre-injection of study intervention on Day 1 and had a normal value of cTnI pre-injection of study intervention on Day 29. Note that other factors such as physical activity can affect cTnI.
Time Frame: Day 4 and Day 32
Population: Evaluable Set: All randomized participants who received at least 1 study injection who had no major protocol deviations or conditions/medications that impacted critical or key analysis data. The 'number of participants analysed' includes the number of participants with normal cTnI at pre-injection at either Day 1 or Day 29 and non-missing cTnI at both pre-injection and 3 days after any injection.
Measure: Count of Participants; unit: Participants
Groups:
- mRNA-1273.712: Participants received mRNA-1273.712 as an IM injection on either Day 1 in Sequence 1 (mRNA-1273.712 - placebo) or Day 29 in Sequence 2 (placebo - mRNA-1273.712) of the study.
- Placebo: Participants received placebo matched to mRNA-1273.712 as an IM injection on either Day 1 in Sequence 2 (placebo - mRNA-1273.712) or Day 29 in Sequence 1 (mRNA-1273.712 - placebo) of the study.
Arm/Group | mRNA-1273.712 | Placebo
Number analyzed (Participants) | 890 | 910
Participants | 1 | 0

2. Secondary Outcome: Number of Participants With Elevated cTnI Level at Day 1 (Baseline)
Description: Elevated cTnI was defined as >53.53 pg/mL in males and >38.64 pg/mL in females.
Time Frame: Pre-injection 1: Day 1
Population: Evaluable Set: All randomized participants who received at least 1 study injection who had no major protocol deviations or conditions/medications that impacted critical or key analysis data. The 'number of participants analysed' includes the number of participants with non-missing cTnI at Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1: mRNA-1273.712 Then Placebo | Sequence 2: Placebo Then mRNA-1273.712
Number analyzed (Participants) | 491 | 489
Participants | 2 | 5

3. Secondary Outcome: Number of Participants With Elevated cTnI Level at Day 29 or Day 57 (28 Days After Injection 1 or Injection 2)
Description: Elevated cTnI was defined as >53.53 pg/mL in males and >38.64 pg/mL in females.
Time Frame: Day 29 and Day 57
Population: Evaluable Set: All randomized participants who received at least 1 study injection who had no major protocol deviations or conditions/medications that impacted critical or key analysis data. The 'number of participants analysed' includes the number of participants with normal cTnI at pre-injection and non-missing cTnI at both pre-injection and 28 days after any injection.
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1273.712 | Placebo
Number analyzed (Participants) | 858 | 853
Participants | 4 | 8

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Medically-attended Adverse Events (MAAEs), Adverse Events of Special Interest (AESIs), and Adverse Events Leading to Withdrawal
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in birth defects or was an important medical event. A MAAE was defined as an AE that led to an unscheduled visit to a healthcare practitioner. Investigators reported AEs as AESIs based on pre-defined criteria. All suspected cases of cardiomyopathy and non-infectious myocarditis, pericarditis, and myopericarditis were reported as AESIs. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Adverse Events' module.
Time Frame: Day 1 up to Day 57
Population: Safety Set: All randomized participants who received at least 1 study injection. Data were collected and presented by study intervention sequence, and treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Sequence 1 (mRNA-1273.712 - Placebo): mRNA-1273.712: Participants received mRNA-1273.712 as an IM injection on Day 1 in Sequence 1 of the study.
- Sequence 1 (mRNA-1273.712 - Placebo): Placebo: Participants received placebo matching mRNA-1273.712 as an IM injection on Day 29 in Sequence 1 of the study.
- Sequence 2 (Placebo - mRNA-1273.712): Placebo: Participants received placebo matched to mRNA-1273.712 as an IM injection on Day 1 in Sequence 2 of the study.
- Sequence 2 (Placebo - mRNA-1273.712): mRNA-1273.712: Participants received mRNA-1273.712 as an IM injection on Day 29 in Sequence 2 of the study.
Arm/Group | Sequence 1 (mRNA-1273.712 - Placebo): mRNA-1273.712 | Sequence 1 (mRNA-1273.712 - Placebo): Placebo | Sequence 2 (Placebo - mRNA-1273.712): Placebo | Sequence 2 (Placebo - mRNA-1273.712): mRNA-1273.712
Number analyzed (Participants) | 500 | 460 | 497 | 454
Participants
  SAEs | 0 | 0 | 0 | 1
  MAAEs | 6 | 5 | 9 | 10
  AESIs | 1 | 1 | 0 | 0
  AEs Leading to Study Discontinuation | 0 | 0 | 1 | 0
  AEs Leading to Discontinuation of Study Injection | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 57
Description: Safety Set: All randomized participants who received at least 1 dose of study injection. Data are presented by study intervention sequence, and treatment received.
Groups:
- mRNA-1273.712 - Placebo Sequence: mRNA-1273.712: Participants received mRNA-1273.712 as an IM injection on Day 1 in Sequence 1 of the study.
- mRNA-1273.712 - Placebo Sequence: Placebo: Participants received placebo matching mRNA-1273.712 as an IM injection on Day 29 in Sequence 1 of the study.
- Placebo - mRNA-1273.712 Sequence: Placebo: Participants received placebo matched to mRNA-1273.712 as an IM injection on Day 1 in Sequence 2 of the study.
- Placebo - mRNA-1273.712: mRNA-1273.712: Participants received mRNA-1273.712 as an IM injection on Day 29 in Sequence 2 of the study.
Arm/Group | mRNA-1273.712 - Placebo Sequence: mRNA-1273.712 | mRNA-1273.712 - Placebo Sequence: Placebo | Placebo - mRNA-1273.712 Sequence: Placebo | Placebo - mRNA-1273.712: mRNA-1273.712
All-Cause Mortality (participants affected / at risk) | 0/500 | 0/460 | 0/497 | 0/454
Serious Adverse Events (participants affected / at risk) | 0/500 | 0/460 | 0/497 | 1/454
Other Adverse Events (participants affected / at risk) | 0/500 | 0/460 | 0/497 | 0/454
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mRNA-1273.712 - Placebo Sequence: mRNA-1273.712 (N=500) | mRNA-1273.712 - Placebo Sequence: Placebo (N=460) | Placebo - mRNA-1273.712 Sequence: Placebo (N=497) | Placebo - mRNA-1273.712: mRNA-1273.712 (N=454)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT06634797/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT06634797/SAP_001.pdf